CLINICAL TRIAL: NCT03066778
Title: A Phase 3 Randomized, Double-Blind, Placebo-controlled Trial of Pembrolizumab (MK-3475/SCH900475) in Combination With Etoposide/Platinum (Cisplatin or Carboplatin) for the First-line Treatment of Subjects With Extensive Stage Small Cell Lung Cancer (KEYNOTE-604)
Brief Title: A Study of Pembrolizumab (MK-3475) in Combination With Etoposide/Platinum (Cisplatin or Carboplatin) for Participants With Extensive Stage Small Cell Lung Cancer (MK-3475-604/KEYNOTE-604)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3475-604; 173744 (Registry Identifier: JAPIC-CTI); MK-3475-604 (Other: Merck); KEYNOTE-604 (Other: Merck); 2016-004309-15 (EudraCT Number)
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Results first posted 2020-12-22 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-08

CONDITIONS: Small Cell Lung Cancer (SCLC)
Keywords: Extensive stage small cell lung cancer (ES-SCLC); Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death Ligand 1 (PDL1, PD-L1); Programmed Cell Death Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Small Cell Lung Carcinoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Saline Solution; Carboplatin; Cisplatin; Etoposide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab+EP (Experimental): During each 21-day cycle, participants receive pembrolizumab 200 mg intravenously (IV) on Day 1 PLUS etoposide 100 mg/m^2 IV on Days 1, 2 and 3 PLUS investigator's choice of platinum therapy (carboplatin titrated to an area under the plasma drug concentration-time curve [AUC] 5 IV on Day 1 OR cisplatin 75 mg/m^2 IV on Day 1). Participants who stop pembrolizumab as a result of obtaining a response of stable disease (SD), partial response (PR), complete response (CR) or those who stop after receiving pembrolizumab for 24 months for reasons other than disease progression or intolerability, are eligible for up to an additional 1 year of treatment after progressive disease if they meet the criteria for retreatment.
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Etoposide
- Placebo+EP (Active Comparator): During each 21-day cycle, participants receive placebo (normal saline solution) IV on Day 1 PLUS etoposide 100 mg/m^2 IV on Days 1, 2 and 3 PLUS investigator's choice of platinum therapy (carboplatin titrated to an AUC 5 IV on Day 1 OR cisplatin 75 mg/m^2 IV on Day 1).
  Interventions: Drug: Normal saline solution; Drug: Carboplatin; Drug: Cisplatin; Drug: Etoposide

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion on Day 1 of each cycle prior to chemotherapy
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab+EP
Drug: Normal saline solution — IV infusion on Day 1 of each cycle prior to chemotherapy
  Arms: Placebo+EP
Drug: Carboplatin — IV infusion on Day 1 of each cycle
  Other Names: PARAPLATIN®
Drug: Cisplatin — IV infusion on Day 1 of each cycle
  Other Names: PLATINOL®
Drug: Etoposide — IV infusion on Days 1, 2 and 3 of each cycle
  Other Names: TOPOSAR™

SUMMARY:
The purpose of this study is to assess the safety and efficacy of pembrolizumab plus standard of care (SOC) chemotherapy (etoposide/platinum [EP]) in participants with newly diagnosed extensive stage small cell lung cancer (ES-SCLC) who have not previously received systemic therapy for this malignancy.

The primary study hypotheses are that pembrolizumab+EP prolongs Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by blinded independent central review (BICR) and Overall Survival (OS) compared with placebo+EP in adult participants with ES-SCLC. In this study, RECIST 1.1 has been modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ.

With protocol Amendment 07 (03-Oct-2018), the outcome measure of "Change from Baseline at Weeks 12 and 24 in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30) Global Health Status/Quality of Life Scale" was replaced with a single time point analysis at Week 18.

ELIGIBILITY:
Inclusion Criteria:

* Has a documented new diagnosis of SCLC by histology or cytology from brushing, washing, or needle aspiration of a defined lesion. Participants who do not have histology samples (defined as core or excisional biopsy, or resections) will need to undergo a new biopsy to provide a tissue sample.
* Has extensive-stage disease defined as Stage IV (T any, N any, M 1a/b) by the American Joint Committee on Cancer (AJCC), Seventh Edition
* Has ≥1 lesion that meets the criteria for measurable, as defined by RECIST 1.1, and is appropriate for selection as a target lesion, as determined by local site investigator/radiology assessment
* Has provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated
* Has Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Has a life expectancy of ≥3 months
* Has adequate organ function
* Female and male participants of childbearing potential must be willing to use an adequate method of contraception, starting with the first dose of study treatment through 120 days after the last dose of study treatment and up to 180 days after last dose of chemotherapeutic agents

Exclusion Criteria:

* Has received prior systemic therapy for the treatment of SCLC
* Is currently participating and receiving study treatment or has participated in a study of an investigational agent and received study treatment or used an investigational device within 4 weeks of the first dose of treatment for another health-related problem
* Is expected to require any other form of antineoplastic therapy for SCLC, including radiation therapy, while on study. (Prophylactic cranial irradiation will be possible for those participants with stable disease or better at the completion of the 4 cycles of chemotherapy with or without pembrolizumab.)
* Has known central nervous system (ie, brain and/or spinal cord) metastases and/or carcinomatous meningitis. Participants with brain metastases may participate only if they satisfy all of the following:
* Has completed treatment (eg, whole brain radiation treatment [WBRT], stereotactic radiosurgery, or equivalent) ≥14 days prior to the first dose of study treatment,
* Has no evidence of new or enlarging brain metastases confirmed by post-treatment repeat brain imaging performed ≥3 weeks after pre-treatment brain imaging, and
* Is neurologically stable without the need for steroids for ≥7 days before first dose of study treatment.
* Has had major surgery within 3 weeks prior to receiving the first dose of study treatment or has not recovered adequately from toxicity and/or complications from an intervention prior to receiving the first dose of study treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has a known history of interstitial lung disease
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include early stage cancers (carcinoma in situ or Stage 1) treated with curative intent, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer, or in situ breast cancer that has undergone potentially curative therapy.
* Has active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy is not considered a form of systemic treatment.
* Has a known history of, or active, neurologic paraneoplastic syndrome
* Has clinically active diverticulitis, intra-abdominal abscess, gastrointestinal obstruction, and/or abdominal carcinomatosis
* Has a history of a severe hypersensitivity reaction to treatment with another monoclonal antibody
* Is taking chronic systemic steroids (in doses exceeding 10 mg daily of prednisone equivalent) within 7 days prior to the first dose of study treatment
* Has a diagnosis of immunodeficiency or is receiving any form of immunosuppressive therapy within 7 days prior to the first dose of study treatment
* Has received a live vaccine within 30 days prior to the first dose of study treatment
* Has received prior therapy with an anti-programmed cell death protein-1 (anti-PD-1), anti-programmed cell death-ligand 1 (anti-PD-L1), or anti-programmed cell death-ligand 2 (anti-PD-L2) agent or with an agent directed to another co-inhibitory T-cell receptor (i.e., cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], tumor necrosis factor receptor superfamily member 9 [TNFRSF9, OX-40, CD137]) or has previously participated in a Merck pembrolizumab (MK-3475) clinical trial
* Has severe hypersensitivity (Grade ≥3) to pembrolizumab and/or any of its excipients
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of Hepatitis B or known active Hepatitis C virus infection
* Has a known history of active TB (Bacillus Tuberculosis)
* Has symptomatic ascites or pleural effusion. A participant who is clinically stable following treatment for these conditions (including therapeutic thoraco- or paracentesis) is eligible.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study starting with the screening visit through 120 days after the last dose of study treatment through and up to 180 days after last dose of chemotherapeutic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2021-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (148):
- United States (27):
  - Baptist Health Medical Group Oncology, LLC ( Site 8000), Miami, Florida
  - Rush University Medical Center ( Site 1215), Chicago, Illinois
  - North Shore University Health System ( Site 1216), Evanston, Illinois
  - Community Hospital ( Site 1207), Munster, Indiana
  - Weinberg Cancer Institute at Franklin Square ( Site 1210), Baltimore, Maryland
  - Massachusetts General Hospital ( Site 1203), Boston, Massachusetts
  - Beth Israel Deaconess Medical Center ( Site 1206), Boston, Massachusetts
  - Dana-Farber Cancer Institute [Boston] ( Site 1201), Boston, Massachusetts
  - University of Michigan ( Site 1217), Ann Arbor, Michigan
  - Henry Ford Health System ( Site 1221), Detroit, Michigan
  - Minnesota Oncology Hematology, PA ( Site 8001), Minneapolis, Minnesota
  - Hattiesburg Clinic ( Site 1205), Hattiesburg, Mississippi
  - Mercy Hospital Saint Louis ( Site 1213), St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada ( Site 8004), Henderson, Nevada
  - Memorial Sloan-Kettering Cancer Center At Basking Ridge ( Site 1226), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center- Monmouth ( Site 1225), Middletown, New Jersey
  - Memorial Sloan-Kettering Cancer Center at Commack ( Site 1227), Commack, New York
  - Memorial Sloan Kettering Cancer Center ( Site 1229), Harrison, New York
  - Memorial Sloan Kettering Cancer Center ( Site 1211), New York, New York
  - Memorial Sloan Kettering Cancer Center - Rockville Centre ( Site 1228), Rockville Centre, New York
  - Montefiore Einstein Center for Cancer Care - Main site ( Site 1204), The Bronx, New York
  - Montefiore Medical Center ( Site 1222), The Bronx, New York
  - Duke University Medical Center ( Site 1214), Durham, North Carolina
  - Bon Secours St. Francis Health Sytem ( Site 1212), Greenville, South Carolina
  - Tennessee Oncology, PLLC/The Sarah Cannon Research Institute ( Site 1230), Nashville, Tennessee
  - Texas Oncology ( Site 8002), Austin, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center ( Site 8003), Dallas, Texas
- Australia (5):
  - Blacktown Hospital ( Site 0004), Blacktown, New South Wales
  - Southern Medical Day Care Centre ( Site 0001), Wollongong, New South Wales
  - St John of God ( Site 0006), Murdoch, Western Australia
  - Lyell McEwin Hospital ( Site 0002), Elizabeth Vale
  - St Vincents Hospital Melbourne ( Site 0005), Fitzroy
- Canada (9):
  - Cancer Care Manitoba ( Site 0159), Winnipeg, Manitoba
  - Nova Scotia Health Authority ( Site 0157), Halifax, Nova Scotia
  - William Osler Health System (Brampton Civic Hospital) ( Site 0161), Brampton, Ontario
  - Kingston Health Sciences Centre ( Site 0155), Kingston, Ontario
  - Sunnybrook Research Institute ( Site 0151), Toronto, Ontario
  - CISSS de la Monteregie-Centre ( Site 0152), Greenfield Park, Quebec
  - CISSS-CA Hotel Dieu de Levis ( Site 0154), Lévis, Quebec
  - CIUSSS Ouest de l'Ile - St-Mary's Hospital ( Site 0158), Montreal, Quebec
  - St. Jerome Medical Research Inc. ( Site 0160), Saint-Jérôme, Quebec
- Chile (5):
  - Instituto Nacional del Cancer ( Site 0207), Santiago, Santiago Metropolitan
  - Health and Care Chile ( Site 0202), Santiago
  - Fundacion Arturo Lopez Perez FALP ( Site 0203), Santiago
  - Pontificia Universidad Catolica de Chile ( Site 0206), Santiago
  - Clinica Universidad Catolica del Maule ( Site 0208), Talca
- France (7):
  - CHRU de Lille - Hopital Albert Calmette ( Site 0353), Lille
  - C.H.R.U. De Limoges ( Site 0358), Limoges
  - CHU Nantes - Hopital Laennec ( Site 0363), Nantes
  - Centre Antoine Lacassagne ( Site 0362), Nice
  - Hopital Tenon ( Site 0360), Paris
  - Institut de Cancerologie Jean-Godinot ( Site 0351), Reims
  - CHU de Toulouse - Hopital Larrey ( Site 0354), Toulouse
- Germany (8):
  - Evangelische Lungenklinik Berlin ( Site 0403), Berlin
  - Medizinische Fakultaet Carl Gustav Carus der TU Dresden ( Site 0411), Dresden
  - Florence Nightingale Krankenhaus ( Site 0413), Düsseldorf
  - SRH Waldklinikum Gera GmbH ( Site 0405), Gera
  - Asklepios Klinikum Harburg ( Site 0412), Hamburg
  - Thoraxklinik Heidelberg gGmbH am Universitaetsklinikum Heidelberg ( Site 0401), Heidelberg
  - Philipps-Universitat Marburg ( Site 0414), Marburg
  - Universitaetsklinikum Tuebingen ( Site 0404), Tübingen
- Hungary (9):
  - Orszagos Onkologiai Intezet ( Site 0453), Budapest, Pest County
  - Orszagos Koranyi TBC es Pulmonologiai Intezet ( Site 0452), Budapest
  - Orszagos Koranyi TBC es Pulmonologiai Intezet ( Site 0458), Budapest
  - Orszagos Koranyi TBC es Pulmonologiai Intezet ( Site 0459), Budapest
  - Veszprem Megyei Tudogyogyintezet ( Site 0454), Farkasgyepű
  - Petz Aladar Megyei Oktato Korhaz ( Site 0460), Győr
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz ( Site 0456), Székesfehérvár
  - Jasz Nagykun Szolnok Megyei Hetenyi Geza Korhaz Rendelointezet ( Site 0451), Szolnok
  - Zala Megyei Szent Rafael Korhaz ( Site 0457), Zalaegerszeg
- Ireland (2):
  - St Vincents University Hospital ( Site 1456), Dublin
  - St James Hospital ( Site 1452), Dublin
- Israel (5):
  - Soroka Medical Center ( Site 0505), Beersheba
  - Ramban Medical Center - Dept. Hemato. & B. Marrow Transplant ( Site 0502), Haifa
  - Meir Medical Center ( Site 0503), Kfar Saba
  - Rabin Medical Center ( Site 0504), Petah Tikva
  - Chaim Sheba Medical Center. ( Site 0501), Ramat Gan
- Japan (16):
  - National Hospital Organization Nagoya Medical Center ( Site 0615), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 0613), Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center ( Site 0614), Matsuyama, Ehime
  - Kurume University Hospital ( Site 0609), Kurume, Fukuoka
  - Hyogo Cancer Center ( Site 0611), Akashi, Hyōgo
  - Kanagawa Cancer Center ( Site 0618), Yokohama, Kanagawa
  - Sendai Kousei Hospital ( Site 0602), Sendai, Miyagi
  - National Hospital Organization Kinki-chuo Chest Medical Center ( Site 0608), Sakai, Osaka
  - Shizuoka Cancer Center Hospital and Research Institute ( Site 0607), Sunto-gun, Shizuoka
  - National Hospital Organization Yamaguchi Ube Medical Center ( Site 0601), Ube, Yamaguchi
  - National Hospital Organization Kyushu Medical Center ( Site 0617), Fukuoka
  - Hiroshima University Hospital ( Site 0604), Hiroshima
  - Niigata Cancer Center Hospital ( Site 0610), Niigata
  - Osaka International Cancer Institute ( Site 0616), Osaka
  - The Cancer Institute Hospital of JFCR ( Site 0606), Tokyo
  - Wakayama Medical University Hospital ( Site 0612), Wakayama
- Canterbury Regional Cancer & Blood Services ( Site 0701), Christchurch, New Zealand
- Poland (9):
  - Mazowiecki Szpital Onkologiczny ( Site 0757), Wieliszew, Masovian Voivodeship
  - Przychodnia Lekarska Komed ( Site 0769), Konin
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II ( Site 0768), Krakow
  - Centrum Onkologii Ziemi Lubelskiej im. sw. Jana z Dukli ( Site 0767), Lublin
  - SKPP UM im. Karola Marcinkowkiego w Poznaniu ( Site 0766), Poznan
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii ( Site 0762), Poznan
  - Wojewodzki Szpital Zespolony im. L. Rydygiera w Toruniu ( Site 0756), Torun
  - Centrum Onkologii-Instytut im. Marii Sklodowskiej-Curie ( Site 0751), Warsaw
  - Dolnoslaskie Centrum Onkologii we Wroclawiu ( Site 0771), Wroclaw
- Russia (5):
  - Belgorod Regional Oncology Dispensary ( Site 0804), Belgorod
  - N.N. Blokhin NMRCO ( Site 0801), Moscow
  - SBI of Stavropol region Pyatigorskiy Oncologic dispensary ( Site 0811), Pyatigorsk
  - SBHI Leningrad Regional Clinical Hospital ( Site 0803), Saint Petersburg
  - Municipal Clinical Oncology Center ( Site 0802), Saint Petersburg
- South Korea (5):
  - Inje University Haeundae Paik Hospital ( Site 0905), Busan
  - National Cancer Center ( Site 0904), Goyang-si
  - Severance Hospital Yonsei University Health System ( Site 0903), Seoul
  - Asan Medical Center ( Site 0901), Seoul
  - Samsung Medical Center ( Site 0902), Seoul
- Spain (8):
  - Hospital Universitario Insular de Gran Canaria ( Site 0952), Las Palmas de Gran Canaria, Gran Canaria
  - Complejo Hospitalario Universitario de A Coruna ( Site 0953), A Coruña
  - Hospital del Mar ( Site 0956), Barcelona
  - Hospital Universitari Vall d Hebron ( Site 0951), Barcelona
  - Hospital Ciudad de Jaen ( Site 0957), Jaén
  - Hospital General Universitario Gregorio Maranon ( Site 0958), Madrid
  - Hospital Universitario Fundacion Jimenez Diaz ( Site 0954), Madrid
  - Hospital Clinico Universitario de Valencia ( Site 0955), Valencia
- Switzerland (3):
  - Kantonsspital Graubuenden ( Site 1403), Chur
  - CHUV Centre Hospitalier Universitaire Vaudois ( Site 1405), Lausanne
  - Universitaetsspital Zuerich ( Site 1404), Zurich
- Taiwan (7):
  - Kaohsiung Chang Gung Memorial Hospital of the C.G.M.F. ( Site 1005), Kaohsiung City
  - China Medical University Hospital. ( Site 1003), Taichung
  - Taichung Veterans General Hospital ( Site 1007), Taichung
  - National Cheng Kung University Hospital ( Site 1004), Tainan
  - Chi Mei Medical Center Liuying ( Site 1006), Tainan
  - National Taiwan University Hospital ( Site 1001), Taipei
  - Taipei Veterans General Hospital ( Site 1002), Taipei
- Turkey (Türkiye) (12):
  - Ege Universitesi Tıp Fakultesi ( Site 1052), Izmir, Bornova
  - Baskent University Adana Dr. Turgut Noyan EAH ( Site 1057), Adana
  - Ankara UTF ( Site 1055), Ankara
  - Hacettepe Universitesi Tip Fakultesi Hastanesi ( Site 1060), Ankara
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji EAH ( Site 1053), Ankara
  - Trakya Uni. Tip Fakultesi ( Site 1063), Edirne
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi ( Site 1058), Istanbul
  - Medipol Hastanesi ( Site 1066), Istanbul
  - Medeniyet Uni. Goztepe Egitim ve Arast. Hast. ( Site 1064), Istanbul
  - Medical Park Izmir Hospital ( Site 1051), Izmir
  - Kocaeli Universitesi Tip Fakultesi ( Site 1061), Kocaeli
  - Inonu Universitesi Tip Fakultesi ( Site 1059), Malatya
- United Kingdom (5):
  - Birmingham Heartlands Hospital ( Site 1162), Birmingham
  - St James s University Hospital ( Site 1161), Leeds
  - North Middlesex Hospital ( Site 1151), London
  - Maidstone Hospital ( Site 1155), Maidstone
  - Mount Vernon Cancer Centre ( Site 1156), Northwood

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Rudin CM, Awad MM, Navarro A, Gottfried M, Peters S, Csoszi T, Cheema PK, Rodriguez-Abreu D, Wollner M, Yang JC, Mazieres J, Orlandi FJ, Luft A, Gumus M, Kato T, Kalemkerian GP, Luo Y, Ebiana V, Pietanza MC, Kim HR; KEYNOTE-604 Investigators. Pembrolizumab or Placebo Plus Etoposide and Platinum as First-Line Therapy for Extensive-Stage Small-Cell Lung Cancer: Randomized, Double-Blind, Phase III KEYNOTE-604 Study. J Clin Oncol. 2020 Jul 20;38(21):2369-2379. doi: 10.1200/JCO.20.00793. Epub 2020 May 29. PMID 32468956
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in the pembrolizumab+ chemotherapy (etoposide/platinum [EP]) arm were eligible to receive second course treatment with pembrolizumab if they met criteria for re-treatment. Per protocol, response, progression, or patient reported outcomes during the second course were not counted towards efficacy outcome measures and adverse events during the second course were not counted towards safety outcome measures.
Pre-assignment Details: One participant who was randomized to the pembrolizumab+EP arm was inadvertently treated with placebo+EP. For efficacy analyses this participant will be included in the arm they were initially randomized into and for safety analyses the participant will be included by treatment received.
Groups:
- Pembrolizumab+EP: During each 21-day cycle, participants received pembrolizumab 200 mg intravenously (IV) on Day 1 PLUS etoposide 100 mg/m^2 IV on Days 1, 2 and 3 PLUS investigator's choice of platinum therapy (carboplatin titrated to an area under the plasma drug concentration-time curve [AUC] 5 IV on Day 1 OR cisplatin 75 mg/m^2 IV on Day 1). Participants who stopped pembrolizumab as a result of obtaining a response of stable disease (SD), partial response (PR), complete response (CR) or those who stopped after receiving pembrolizumab for 24 months for reasons other than disease progression or intolerability, were eligible for up to an additional 1 year of treatment after progressive disease if they met the criteria for retreatment.
- Placebo+EP: During each 21-day cycle, participants received placebo (normal saline solution) IV on Day 1 PLUS etoposide 100 mg/m^2 IV on Days 1, 2 and 3 PLUS investigator's choice of platinum therapy (carboplatin titrated to an AUC 5 IV on Day 1 OR cisplatin 75 mg/m^2 IV on Day 1).
Period: Overall Study
Arm/Group | Pembrolizumab+EP | Placebo+EP
Started | 228 | 225
Treated | 223 (1 participant randomized to the pembrolizumab+EP arm was treated with placebo+EP.) | 223
Received Second Course of Pembrolizumab | 1 | 0
Completed | 28 | 13
Not Completed | 200 | 212
Not completed — Death | 195 | 205
Not completed — Withdrawal by Subject | 5 | 7

BASELINE CHARACTERISTICS:
Population: All participants randomized by intention to treat (ITT).
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab+EP | Placebo+EP | Total
Number analyzed (Participants) | 228 | 225 | 453
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.2 (8.4) | 65.2 (8.2) | 64.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 83 | 159
  Male | 152 | 142 | 294
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 13 | 19
  Not Hispanic or Latino | 204 | 192 | 396
  Unknown or Not Reported | 18 | 20 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 52 | 34 | 86
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 162 | 177 | 339
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 13 | 13 | 26
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — An ECOG Performance Status of 0 (Fully active, able to carry on all pre-disease performance without restriction) or 1 (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature) was required for inclusion in the study and randomization was stratified by ECOG score.
  Participants
    ECOG = 0 | 60 | 56 | 116
    ECOG = 1 | 168 | 169 | 337
Lactate Dehydrogenase (LDH) Status at Baseline [Count of Participants; unit: Participants] — Randomization of participants in the study was stratified by LDH measurement at baseline ( ≤ or > upper limit of normal).
  Participants
    LDH = ≤ Upper Limit of Normal | 100 | 95 | 195
    LDH = > Upper Limit of Normal | 127 | 129 | 256
    LDH Result Missing | 1 | 1 | 2
Platinum Therapy Administered [Count of Participants; unit: Participants] — Randomization of participants was stratified by type of platinum therapy administered during the study.
  Participants
    Cisplatin | 63 | 66 | 129
    Carboplatin | 161 | 156 | 317
    Not Treated with Platinum Therapy | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. PD, as determined by RECIST 1.1, was defined as ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. For this study, RECIST 1.1 was modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. The PFS was calculated using the non-parametric Kaplan-Meier method for censored data and presented for the first course of study treatment per protocol.
Time Frame: Up to approximately 30.5 months
Population: The analysis population consisted of all randomized participants who were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+EP | Placebo+EP
Number analyzed (Participants) | 228 | 225
Months | 4.8 [4.3 to 5.4] | 4.3 [4.2 to 4.5]
Statistical Analysis 1: Comparison: Pembrolizumab+EP vs Placebo+EP; Test type: Superiority; p = 0.00069, Log Rank; One-sided p-value based on log-rank test stratified by platinum chemotherapy, ECOG, and LDH; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.60 to 0.88] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by platinum chemotherapy, ECOG, and LDH

2. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the analysis were censored at the date of the last follow up. The OS was calculated using the non-parametric Kaplan-Meier method for censored data and presented for the first course of study treatment per protocol.
Time Frame: Up to approximately 30.5 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+EP | Placebo+EP
Number analyzed (Participants) | 228 | 225
Months | 10.8 [9.2 to 12.9] | 9.7 [8.6 to 10.7]
Statistical Analysis 1: Comparison: Pembrolizumab+EP vs Placebo+EP; Test type: Superiority; p = 0.01643, Log Rank; One-sided p-value based on log-rank test stratified by platinum chemotherapy, ECOG, and LDH; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.64 to 0.98] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: ORR was defined as the percentage of participants who achieve a best objective response of complete response (CR) or partial response (PR) per RECIST 1.1. CR was defined as the disappearance of all target lesions. PR was defined as ≥30% decrease in the sum of diameters of target lesions taking as a reference the baseline sum diameters. In this study, RECIST 1.1 was modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. The ORR was calculated using the Miettinen & Nurminen method stratified by type of platinum therapy (carboplatin or cisplatin), baseline ECOG performance status (0 or 1), and baseline LDH (≤ or > upper limit of normal) and presented for the first course of study treatment per protocol.
Time Frame: Up to approximately 30.5 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab+EP | Placebo+EP
Number analyzed (Participants) | 228 | 225
Percentage of Participants | 70.6 [64.2 to 76.4] | 61.8 [55.1 to 68.2]
Statistical Analysis 1: Comparison: Pembrolizumab+EP vs Placebo+EP; Test type: Superiority; p = 0.02270, Miettinen & Nurminen; One-sided p-value for testing. H0: difference in percent = 0 versus H1: difference in percent > 0; Percent Difference = 8.9, 95% CI 2-sided [0.2 to 17.4] — Based on Miettinen & Nurminen method stratified by platinum chemotherapy, ECOG, and LDH. Cisplatin, ECOG 0, LDH ≤ULN and Cisplatin, ECOG 0, LDH >ULN were combined into one stratum because of small sample size

4. Secondary Outcome: Duration of Response (DOR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: DOR was defined as the time from first documented evidence of a Complete Response (CR) or Partial Response (PR) per RECIST 1.1 until progressive disease (PD) per RECIST 1.1 or death due to any cause, whichever occurred first. CR was defined as the disappearance of all target lesions. PR was defined as ≥30% decrease in the sum of diameters of target lesions taking as a reference the baseline sum diameters. PD was defined as ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of ≥1 new lesions was also considered PD. In this study, RECIST 1.1 was modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. The DOR was calculated using the product-limit (Kaplan-Meier) method for censored data and is presented for the first course of study treatment per protocol.
Time Frame: Up to approximately 30.5 months
Population: The analysis population consisted of all randomized participants who were included in the treatment group to which they were randomized and experienced a CR or PR.
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab+EP | Placebo+EP
Number analyzed (Participants) | 161 | 139
Months | NA [NA to NA] — NA=median DOR and upper and lower limits not reached due to no progressive disease by time of last disease assessment | NA [NA to NA] — NA=median DOR and upper and lower limits not reached due to no progressive disease by time of last disease assessment

5. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An adverse event was defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which did not necessarily have to have had a causal relationship with this treatment. An adverse event could therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that was temporally associated with the use of the Sponsor's product, was also an adverse event. The number of participants who experienced an AE was reported for each arm according to the treatment received and is presented for the first course of study treatment per protocol.
Time Frame: Up to approximately 30.5 months
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab+EP | Placebo+EP
Number analyzed (Participants) | 223 | 223
Participants | 223 | 222

6. Secondary Outcome: Number of Participants Discontinuing Study Treatment Due to an Adverse Event (AE)
Description: An adverse event was defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which did not necessarily have to have had a causal relationship with this treatment. An adverse event could therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that was temporally associated with the use of the Sponsor's product, was also an adverse event. The number of participants who discontinued due to an AE was reported for each arm according to the treatment received and is presented for the first course of study treatment per protocol.
Time Frame: Up to approximately 26 months
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab+EP | Placebo+EP
Number analyzed (Participants) | 223 | 223
Participants | 33 | 14

7. Secondary Outcome: Number of Participants Experiencing Any Grade 3 to 5 Adverse Events (AE) as Assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events Version 4.03 (CTCAE 4.03)
Description: The CTCAE uses Grades 1 through 5 correlating to AE severity criteria. Grade 1=mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2=moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3=severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4=life-threatening consequences; urgent intervention indicated. Grade 5=death related to AE. The number of participants who experienced any Grade 3 to 5 AE was reported for each arm according to the treatment received and is presented for the first course of study treatment per protocol.
Time Frame: Up to approximately 30.5 months
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab+EP | Placebo+EP
Number analyzed (Participants) | 223 | 223
Participants | 175 | 172

8. Secondary Outcome: Change From Baseline at Week 18 in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30) Global Health Status/Quality of Life Scale
Description: EORTC QLQ-C30 is a questionnaire that rates the overall quality of life in cancer participants. The first 28 questions use a 4-point scale (1=not at all to 4=very much) for evaluating function (physical, role, social, cognitive, emotional), symptoms (diarrhea, fatigue, dyspnea, appetite loss, insomnia, nausea/vomiting, constipation, and pain) and financial difficulties. The last 2 questions use a 7-point scale (1=very poor to 7=excellent) to evaluate overall health and quality of life. Scores are transformed to a range of 0 to 100 using a standard EORTC algorithm. Change from baseline scores were calculated using a constrained longitudinal data analysis (cLDA) model. Negative change from baseline values indicated deterioration in health status or functioning and positive changes indicated improvement. Data are presented for the first course of study treatment per protocol.
Time Frame: Baseline (prior to first dose of study treatment in Cycle 1 [cycle length = 21 days]) and Week 18
Population: All participants who received at least 1 dose of study medication and had non-missing assessments at baseline and Week 18.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab+EP | Placebo+EP
Number analyzed (Participants) | 221 | 218
Score on a Scale | 8.66 [5.26 to 12.06] | 4.23 [0.93 to 7.52]
Statistical Analysis 1: Comparison: Pembrolizumab+EP vs Placebo+EP; Test type: Other; p = 0.040, Log Rank; Difference in Least Square Means = 4.43, 95% CI 2-sided [0.21 to 8.66]

9. Secondary Outcome: Change From Baseline at Week 12 in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30) Global Health Status/Quality of Life Scale
Description: EORTC QLQ-C30 is a questionnaire that rates the overall quality of life in cancer participants. The first 28 questions use a 4-point scale (1=not at all to 4=very much) for evaluating function (physical, role, social, cognitive, emotional), symptoms (diarrhea, fatigue, dyspnea, appetite loss, insomnia, nausea/vomiting, constipation, and pain) and financial difficulties. The last 2 questions use a 7-point scale (1=very poor to 7=excellent) to evaluate overall health and quality of life. Scores were transformed to a range of 0 to 100 using a standard EORTC algorithm. Negative change from baseline values indicated deterioration in health status or functioning and positive changes indicated improvement. Per protocol, data were to be presented for the first course of study treatment.
Time Frame: Baseline (prior to first dose of study treatment in Cycle 1 [cycle length = 21 days]) and Week 12
Population: All participants who received at least 1 dose of study medication and had non-missing assessments at baseline and Week 12. This outcome measure was replaced with a single time-point analysis at Week 18 as pre-specified with Amendment 7 of the protocol (03-Oct-2018).
Arm/Group | Pembrolizumab+EP | Placebo+EP
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline at Week 24 in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30) Global Health Status/Quality of Life Scale
Description: as for outcome 9
Time Frame: Baseline (prior to first dose of study treatment in Cycle 1 [cycle length = 21 days]) and Week 24
Population: All participants who received at least 1 dose of study medication and had non-missing assessments at baseline and Week 24. This outcome measure was replaced with a single time-point analysis at Week 18 as pre-specified with Amendment 7 of the protocol (03-Oct-2018).
Arm/Group | Pembrolizumab+EP | Placebo+EP
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Time to True Deterioration (TTD) in the Composite Endpoint of Cough, Chest Pain, and Dyspnea Using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30) and Lung Cancer Module 13 (QLQ-LC13)
Description: TTD in patient-reported lung cancer symptoms of cough (QLQ-LC-13 Item 1), chest pain (QLQ-LC-13 Item 10), and dyspnea (QLQ-C30 Item 8) was a composite endpoint defined as the time to first onset of ≥10 point deterioration from baseline in an item confirmed by a second adjacent ≥10 point deterioration. The QLQ-LC13 consists of 13 measures of lung cancer symptoms and side effects from chemotherapy and radiation. It is scored on a 4-point scale (1=none, 2=a little, 3=quite a bit, 4=very much). Scores were transformed to a range of 0 to 100 using a standard algorithm. Higher scores represented increasing symptom severity. TTD was calculated using the product-limit Kaplan-Meier method for censored data and is presented for the first course of study treatment per protocol.
Time Frame: Day 1 of Cycles 1-9, Day 1 of every other cycle for Cycles 10-17 and 30 days after last dose of study treatment (Up to approximately 27 months)
Population: All participants who received at least 1 dose of study medication and had non-missing assessments.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+EP | Placebo+EP
Number analyzed (Participants) | 221 | 218
Months | NA [NA to NA] — Median TTD and lower and upper limits not reached (no protocol-specified deterioration criteria reached by time of last assessment) | 8.7 [5.9 to NA] — TTD upper limit not reached (no protocol-specified deterioration criteria reached by time of last assessment)
Statistical Analysis 1: Comparison: Pembrolizumab+EP vs Placebo+EP; Test type: Other; p = 0.208, Log Rank; Two-sided p-value based on stratified log-rank test; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.56 to 1.14] — Based on Cox regression model with treatment as a covariate stratified by platinum chemotherapy ECOG, and LDH. Cisplatin, ECOG 0, LDH ≤ULN and Cisplatin, ECOG 0, LDH >ULN were combined into one stratum because of small sample size

ADVERSE EVENTS:
Time Frame: First Course: Up to 49.5 months Second Course: Up to 37.9 months First and second course dosing occurred concurrently
Description: All-cause mortality (ACM)=all randomized participants; AE=all participants who received ≥1 dose of study treatment. Per protocol, MedDRA preferred terms neoplasm progression (NP), malignant NP, disease progression not related to study treatment are excluded. ACM was adjusted for the participant who was randomized to pembrolizumab+EP and treated with placebo+EP. AEs presented by actual treatment received. Per protocol, collection of AE and ACM were planned for first and second courses.
Groups:
- Pembrolizumab Second Course: Participants who met the criteria for retreatment received pembrolizumab 200 mg by IV infusion on Day 1 of each 21-day cycle for up to 1 year of treatment.
Arm/Group | Pembrolizumab+EP | Placebo+EP | Pembrolizumab Second Course
All-Cause Mortality (participants affected / at risk) | 196/227 | 212/226 | 1/1
Serious Adverse Events (participants affected / at risk) | 111/223 | 89/223 | 1/1
Other Adverse Events (participants affected / at risk) | 221/223 | 216/223 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab+EP (N=223) | Placebo+EP (N=223) | Pembrolizumab Second Course (N=1)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 10 (10) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 15 (15) | 14 (14) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 11 (11) | 6 (6) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 5 (6) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 3 (3) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Autoimmune uveitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 3 (3) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 4 (4) | 3 (3) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Paracancerous pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pleural infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 17 (20) | 12 (13) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Serratia sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (6) | 5 (11) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Limbic encephalitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (7) | 1 (1) | 0 (0)
Autoimmune nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Neurogenic bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Subacute cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab+EP (N=223) | Placebo+EP (N=223) | Pembrolizumab Second Course (N=1)
Anaemia (Blood and lymphatic system disorders) | 101 (122) | 96 (115) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 49 (84) | 45 (70) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 120 (217) | 114 (207) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 57 (85) | 46 (80) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 12 (12) | 6 (7) | 0 (0)
Hypothyroidism (Endocrine disorders) | 26 (27) | 5 (5) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 15 (18) | 13 (13) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 13 (14) | 5 (5) | 0 (0)
Constipation (Gastrointestinal disorders) | 65 (78) | 59 (69) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 46 (67) | 41 (48) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 12 (13) | 7 (7) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 12 (12) | 6 (6) | 0 (0)
Nausea (Gastrointestinal disorders) | 85 (135) | 96 (144) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 14 (17) | 15 (17) | 0 (0)
Vomiting (Gastrointestinal disorders) | 36 (48) | 39 (49) | 0 (0)
Asthenia (General disorders) | 38 (46) | 43 (48) | 0 (0)
Chest pain (General disorders) | 11 (11) | 21 (24) | 0 (0)
Fatigue (General disorders) | 61 (76) | 60 (78) | 0 (0)
Oedema peripheral (General disorders) | 17 (20) | 26 (32) | 0 (0)
Pyrexia (General disorders) | 32 (37) | 14 (17) | 0 (0)
Nasopharyngitis (Infections and infestations) | 12 (15) | 9 (9) | 0 (0)
Pneumonia (Infections and infestations) | 12 (13) | 13 (14) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 17 (22) | 13 (16) | 0 (0)
Urinary tract infection (Infections and infestations) | 10 (12) | 8 (9) | 1 (1)
Alanine aminotransferase increased (Investigations) | 17 (20) | 21 (24) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 19 (22) | 13 (15) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 12 (15) | 6 (8) | 0 (0)
Blood creatinine increased (Investigations) | 15 (23) | 8 (8) | 0 (0)
Weight decreased (Investigations) | 22 (24) | 20 (23) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 69 (85) | 54 (68) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 15 (20) | 13 (19) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 21 (26) | 16 (23) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 (37) | 19 (22) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 25 (27) | 26 (27) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 12 (14) | 6 (6) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (15) | 13 (16) | 0 (0)
Dizziness (Nervous system disorders) | 31 (36) | 15 (17) | 0 (0)
Dysgeusia (Nervous system disorders) | 14 (14) | 12 (13) | 0 (0)
Headache (Nervous system disorders) | 29 (34) | 34 (41) | 0 (0)
Insomnia (Psychiatric disorders) | 25 (26) | 28 (34) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 45 (62) | 45 (51) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 37 (41) | 37 (41) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 75 (77) | 84 (87) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 13 (13) | 10 (10) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 13 (14) | 4 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 25 (33) | 18 (23) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 30 (39) | 13 (17) | 0 (0)
Hypertension (Vascular disorders) | 12 (15) | 10 (14) | 0 (0)
Hypotension (Vascular disorders) | 9 (11) | 16 (21) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/78/NCT03066778/Prot_SAP_001.pdf